

# BROWN UNIVERSITY CONSENT FOR RESEARCH PARTICIPATION

Version 1 06/22//2023

Study Title: Developing and Testing a Produce Prescription Implementation blueprint to improve food security in a clinical setting: A pilot study

You are invited to take part in a Brown University research study. Your participation is voluntary.

RESEARCHERS: **Alison Tovar, PhD, MPH** (alison\_tovar@brown.edu, 401-863-7327) & **Hannah Frank, PhD** (hannah frank@brown.edu, 401-444-1941).

PURPOSE: The vegetable program that you are participating in is trying some additional ways to improve the program and we are testing how well these work.

PROCEDURES: You will be asked to participate in surveys at the start and end of the vegetable program season, which is about six months. You will also receive a very brief (4 question) biweekly text or phone call survey. After the final delivery, at six months, you will complete a similar survey to the one you completed at the beginning.

TIME INVOLVED: The surveys given at the beginning and after the final delivery are expected to take about 15-20 minutes of your time. The biweekly surveys are expected to take 1-2 minutes of your time. The study period lasts six months.

COMPENSATION: After completing the survey measures, you will be given a \$50 gift card for your time during the initial survey. For the biweekly questions, you will be given \$3 for each survey you answer. After the final surveys are completed, you will be given \$75 and the total amount corresponding to the number of biweekly surveys that you completed. You could be given up to a total of approximately \$164 for your participation in the study.

RISKS: You may be uncomfortable answering questions about your experience with the vegetable program, people involved in it, or access to food. You do not have to answer

any questions you do not want to on the surveys. Leaving the study will not affect your relationship with Brown University or the vegetable program.

BENEFITS: Although there is not a direct benefit to you. You potentially can improve the vegetable program for families who participate in the future.

CONFIDENTIALITY: Information that may be used to identify you will only be documented on consent forms and contact information forms. Your survey responses will be assigned a number that has no association with your identity to protect your responses. No personally identifiable information will be collected in the survey. All contact information will be stored in a private Google Drive that is only accessible to study personnel. This information will only be used for scheduling and compensation purposes and will be deleted 30 days after you complete the final survey. Electronic consent forms will be stored on the Qualtrics platform, and access to these forms will be limited to research personnel. These forms will be stored for three years after the study has ended, and then destroyed.

Brown University Institutional Review Board sometimes reviews studies like this one to make sure they are being done safely and correctly. If a review of this study takes place, your records may be examined. The researchers will protect your confidentiality.

A description of this study will be available on http://www.ClinicalTrials.gov. This website will not include information that can identify you and if any data is presented, it will only be a summary of the results with no identifiable information. You can search this website at any time.

When the study is finished, researchers will write reports and present what they learned. These reports and presentations will not list your name. No one will know you were in the study unless you tell them. Researchers will also put some of the reports on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>. This website will not include information that can identify you.

VOLUNTARY: You do not have to be in this study if you do not want to be. Even if you decide to be in this study, you can change your mind and stop at any time.

CONTACT INFORMATION: If you have any questions about your participation in this study, you can call **Alison Tovar** at 401-863-7327 or email alison\_tovar@brown.edu, or **Hannah Frank** at 401-444-1941 or email hannah\_frank@brown.edu.

YOUR RIGHTS: If you have questions about your rights as a research participant, you can contact Brown University's Human Research Protection Program at 401-863-3050 or email them at IRB@Brown.edu.

#### CONSENT TO PARTICIPATE

Circle or Click "Yes" or "No" for each statement below:

| • | Do you agree to and understand the information in this document? | Yes |
|---|---|---|
| | No | |
| • | Do you agree to volunteer as a research participant for this study? | Yes |
| | No | |
| ٠ | Would you like a copy of this form with your signature? | Yes |
| | No | |

# If in person

Your signature below shows that you have read and understood the information in this document, and that you agree to volunteer as a research participant for this study.

Participant's Signature and Date / PRINTED NAME

You will be offered a copy of your signed consent form.

#### If electronically

By clicking "Agree" it shows that you have read and understood the information in this document, and that you agree to volunteer as a research participant for this study.



#### **BROWN UNIVERSITY**

## CONSENT FOR RESEARCH PARTICIPATION FOR HEALTHCARE PROVIDERS

Version 2 6/22/2023

Study Title: Developing and Testing a Produce Prescription Implementation blueprint to improve food security in a clinical setting: A pilot study

You are invited to take part in a Brown University research study. Your participation is voluntary.

RESEARCHERS: **Alison Tovar, PhD, MPH** (alison\_tovar@brown.edu, 401-863-7327) & **Hannah Frank, PhD** (hannah frank@brown.edu, 401-444-1941).

PURPOSE: The vegetable program that you are referring patients to is trying some additional ways to improve the program and we are testing how well these work for both patients and for healthcare providers/staff that refer patients.

PROCEDURES: You will be asked to complete one 10-20 minute survey at the beginning before the program begins, and one survey after the program has ended after approximately 6 months.

TIME INVOLVED: The surveys given at the baseline assessments and final study assessments are expected to take about 10-20 minutes of your time.

COMPENSATION: After completing the baseline survey measures, you will be given a \$50 gift card for your time. After the final surveys, you will be given a \$75 gift card. You will be given a total of \$125 for your participation and completing all the surveys in the study.

RISKS: You may be uncomfortable answering questions about your experience with the vegetable program, people involved in it, or access to food. You do not have to answer any questions you do not want to on the surveys. Leaving the study will not affect your relationship with Brown University or the vegetable program.

BENEFITS: Although there is not a direct benefit to you. You potentially can improve the vegetable program for families who participate in the future.

CONFIDENTIALITY: Information that may be used to identify you will only be documented on consent forms and contact information forms. Your survey responses will be assigned a number that has no association with your identity to protect your responses. No personally identifiable information will be collected in the survey. All contact information will be stored in a private Google Drive that is only accessible to study personnel. This information will only be used for scheduling and compensation purposes and will be deleted 30 days after you complete the final survey. Electronic consent forms will be stored on the Qualtrics platform, and access to these forms will be limited to research personnel. These forms will be stored for three years after the study has ended, and then destroyed.

Brown University Institutional Review Board sometimes reviews studies like this one to make sure they are being done safely and correctly. If a review of this study takes place, your records may be examined. The researchers will protect your confidentiality.

A description of this study will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

When the study is finished, researchers will write reports and present what they learned. These reports and presentations will not list your name. No one will know you were in the study unless you tell them. Researchers will also put some of the reports on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>. This website will not include information that can identify you.

VOLUNTARY: You do not have to be in this study if you do not want to be. Even if you decide to be in this study, you can change your mind and stop at any time.

CONTACT INFORMATION: If you have any questions about your participation in this study, you can call **Alison Tovar** at 401-863-7327 or email alison\_tovar@brown.edu, or **Hannah Frank** at 401-444-1941 or email hannah frank@brown.edu.

YOUR RIGHTS: If you have questions about your rights as a research participant, you can contact Brown University's Human Research Protection Program at 401-863-3050 or email them at IRB@Brown.edu.

#### CONSENT TO PARTICIPATE

| Circle "Yes" | or "No" for each statement below: | |
|---|---|---|
| • | Do you agree to and understand the information in this document? | Yes |
| | No | |
| • | Do you agree to volunteer as a research participant for this study? | Yes |
| | No | |

Would you like a copy of this form with your signature? Yes No

# If in person

Your signature below shows that you have read and understood the information in this document, and that you agree to volunteer as a research participant for this study.

Participant's Signature and Date / PRINTED NAME

You will be offered a copy of your signed consent form.

### If electronically

By clicking "Agree" you acknowledge to have read and understood the information in this document, and that you agree to volunteer as a research participant for this study.